CLINICAL TRIAL: NCT03590548
Title: Assiut University Children 's Hospital
Brief Title: Clinical Audit of Managment of Gausher Disease in Children
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Yasmeen Abd Elbaset Hamzaa (Other)
Responsible Party: Sponsor-Investigator, Yasmeen Abd Elbaset Hamzaa, Assiut University, Assiut University
Organization: Assiut University (Other)
Other Study IDs: egypt AssiutU
Record Dates: First submitted 2018-07-07; First posted 2018-07-18 (Actual); Last update posted 2018-07-18 (Actual); Status verified 2018-07

CONDITIONS: Gaucher Disease
MeSH Terms: conditions — Gaucher Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- gausher disease in children: • Inclusion criteria: All cases with confirmed diagnosis of Gaucher disease type 1 and type 3 receiving enzyme replacement therapy at Assuit University Children's Hospital.
  Interventions: Diagnostic Test: gausher disease

INTERVENTIONS:
Diagnostic Test: gausher disease — lab investigation and radio logical

SUMMARY:
clinical audit on managment of gausher disease in children

DETAILED DESCRIPTION:
The main aim of study is to evaluate the management of Gausher disease patient under enzyme replacement therapy in Assuit University Children's Hospital and compare our policy for management with International guideline of management of Gausher disease in children (8)

* Type of study : clinical audit
* Inclusion criteria: All cases with confirmed diagnosis of Gaucher disease type 1 and type 3 receiving enzyme replacement therapy at Assuit University Children's Hospital.
* Site of study :Assuit University children's Hospital Methodiological
* Exclusion criteria 3-New diagnosed cases not on ERT. 2-other lipid storage disease.
* Patient& method The study will include 42 diagnosed Gaucher disease patient under enzyme replacement therapy attend the hematology unit in Assuit University Children's Hospital in one year Reviewing the proposal will be carried out before starting via the ethical committee of Assuit Faculty of Medicine.
* Ethical consideration The aim of the study will be explained to each patient before beginning of the process.

We will compare our policy in management of Gausher disease with International guideline of management of gausher disease

1-cases of Gaucher type 2.

ELIGIBILITY:
Inclusion Criteria:

* All cases with confirmed diagnosis of Gaucher disease type 1 and type 3 receiving enzyme replacement therapy at Assuit University Children's Hospital.

Exclusion Criteria:

* 1-cases of Gaucher type 2. 2-other lipid storage disease. 3-New diagnosed cases not on ERT.

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study will include 42 diagnosed Gaucher disease patient under enzyme replacement therapy attend the hematology unit in Assuit University Children's Hospital in one year
Sampling Method: Non-Probability Sample
Enrollment: 1 (Estimated)
Dates: Start 2018-07 (Estimated); Primary Completion 2018-12 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
evaluate the management of Gausher disease patient under enzyme replacement therapy in Assuit University Children's Hospital and compare our policy for management with International guideline of management of Gausher disease in children (8) | one year
  • Type of study : clinical audit

CONTACTS AND LOCATIONS:
Overall Officials: Mervit Amin, doctora, Principal Investigator — Assiut unversity

IPD SHARING:
Plan to Share IPD: No